CLINICAL TRIAL: NCT06690944
Title: Physical Functioning Adaptations Following a Resisted Functional Exercise Program Based on the Proprioceptive Neuromuscular Facilitation Concept in Older Individuals: a Randomized Clinical Trial
Brief Title: Exercise Based on Proprioceptive Neuromuscular Facilitation in Older Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Eduardo Lusa Cadore, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URioGrandePNF
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Functional Disability; Dynapenia; Sarcopenia in Elderly
Keywords: Frailty; Proprioceptive Neuromuscular Facilitation; Gait; Balance; Sit-Stand; Functionality
MeSH Terms: conditions — Frailty | interventions — Muscle Stretching Exercises; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation Group (Experimental): The Proprioceptive Neuromuscular Facilitation group (PNFG) intervention consisted of applying PNF concept exercises and techniques related to facilitating sitting and walking, carried out by a therapist with basic IPNFA® (International Proprioceptive Neuromuscular Facilitation Association) instruction. The PNF intervention was divided into two stages: Stage 1: which consisted of facilitating stability and controlled mobility of the initial position and phases 1, 2, 3, of the sit-up. At the initial position, we applied PNF stabilizing reversals technique for 2 minutes, to stimulate stability in the upright sitting position. In phase 1, we applied PNF to stimulate controlled mobility of the anterior inclination of the erect trunk. In Phase 2, to improve the concentric and eccentric control of lower limb extensor muscles and, in Phase 3 to improve the stability in an upright position again. Stage 2: consists of facilitating activities related to gait.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation
- Physical exercise without proprioceptive neuromuscular facilitation control group (Active Comparator): The physical exercise without proprioceptive neuromuscular facilitation control group (CG) Intervention consisted of the same activities carried out in the proprioceptive neuromuscular facilitation group (PNFG) during Stages 1 and 2, during the same amount of minutes, sessions, and weeks; however, CG intervention did not include specific techniques and basic principles (i.e. approximation and optimal resistance) and procedures of the PNF concept. The activities were instructed and supervised by a trained professional through verbal command. The professional was at stand-by assistant position to prevent accidents.
  Interventions: Other: Physical exercise without proprioceptive neuromuscular facilitation control group

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — The following basic principles and procedures were emphasized when applying the techniques: manual contact, resistance, approximation, verbal commands, and therapist's body mechanics. During stages 1 and 2 of the intervention, the amount of PNF optimal resistance used was necessary to maintain a stable and safe position, with good body alignment, in a manner that produced coordinated movements to generate appropriate motor learning.
  Arms: Proprioceptive Neuromuscular Facilitation Group
Other: Physical exercise without proprioceptive neuromuscular facilitation control group — The physical exercise without proprioceptive neuromuscular facilitation control group (CG) intervention consisted of the same activities carried out in the proprioceptive neuromuscular facilitation (PNF) group during Stages 1 and 2, during the same amount of minutes, sessions, and weeks; however, CG intervention did not include specific techniques and basic principles (i.e. approximation and optimal resistance) and procedures of the PNF concept. The activities were instructed and supervised by a trained professional through verbal command. The professional was at stand-by assistant position to prevent accidents.
  Arms: Physical exercise without proprioceptive neuromuscular facilitation control group

SUMMARY:
The goal of this clinical trial was to determine whether an intervention using resisted sit-to-stand and walking exercises with Proprioceptive Neuromuscular Facilitation (PNF) techniques improved gait and sit-to-stand in older individuals with poor functional capacity compared to a control group that performed the same activities, but without manual resistance. The main questions it aimed to answer were:

Did an exercise program based on the PNF concept improve functional capacity and strength performance?

Was there a difference between an exercise program with or without PNF techniques on functional capacity and strength in older adults?

Researchers compared the effects of an exercise program based on the PNF concept to a similar exercise training without manual resistance on functional capacity and strength performance.

Participants participated in an intervention using resisted sit-to-stand and walking exercises with or without PNF and performed functional capacity and strength tests at the beginning and end of the intervention.

DETAILED DESCRIPTION:
The proposal consisted of investigating an exercise intervention based on the Proprioceptive Neuromuscular Facilitation concept (PFNG), compared to a control group (CG), which performed the same exercises as PNFG under a therapist's supervision, but without resistance imposed by the therapist's hands as in PFNG, in older individuals.

Before data collection, individuals participated in a familiarization procedure for each test. Each specific test was conducted on the same equipment with identical participant/equipment positioning. Functional assessment and intervention were conducted at the participants' residences.

The CG intervention consisted of the same activities carried out in the PNFG during Stages 1 and 2, for the same amount of minutes, sessions, and weeks. However, the CG intervention did not include specific techniques and basic principles (i.e., approximation and optimal resistance) and procedures of the PNF concept. The activities were instructed and supervised by a trained professional through verbal commands. The professional was in a stand-by assistant position to prevent accidents. Each intervention lasted 30 minutes and took place twice a week, for 4 weeks, totaling 8 meetings. The interventions were supervised by researchers blinded to pre-intervention assessment results and randomly assigned for both PNF and control groups. The researchers responsible for the interventions were physical therapists with basic IPNFA® (International Proprioceptive Neuromuscular Facilitation Association) instruction.

ELIGIBILITY:
Inclusion Criteria:

* Short Physical Performance Battery score lower than 10 points.

Exclusion Criteria:

* Neurodegenerative diseases;
* Illnesses contraindicating exercise (e.g., uncontrolled arrhythmias, acute myocardial infarction);
* Unstable medical condition.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Baseline and immediately after the intervention
  Short Physical Performance Battery (SPPB) includes usual walking speed over 4 meters, balance, and five times sit-to-stand. The sum of the three individual categorical scores yielded the final SPPB score, which ranged from 0 (worst) to 12 (best).

SECONDARY OUTCOMES:
Timed Up and Go | Baseline and immediately after the intervention
  The Timed Up and Go test consists of measuring the time required to perform the task of standing from a chair, walking 3 meters, turning, going back, and sitting down on the chair.
Handgrip strength | Baseline and immediately after the intervention
  Handgrip strength is measured using a hand dynamometer (Jamar Hydraulic Hand Dynamometer). The dynamometer is squeezed twice with each hand while the participant is seated. The upper arm is positioned close to the body with the elbow at a 90° angle. The higher score is used, provided the difference does not exceed 10%; otherwise, a third measurement is taken.
Gait speed | Baseline and immediately after the intervention
  Gait speed is assessed through a 4-meter walking test. Participants are asked to walk 4 meters at their usual speed on a horizontal walkway.
Static balance | Baseline and immediately after the intervention
  Static balance is assessed through 10-second hold parallel feet, semi-tandem, and tandem positions. Participants progress to the hardest test only if they succeed in the easiest.
Sit-To-Stand | Baseline and immediately after the intervention
  The sit-to-stand test consists of the time spent standing from a chair 5 times.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola de Educação Física Fisioterapia e Dança - UFRGS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the end of the study, no end date for sharing IPD was set.
Access Criteria: Researchers affiliated with recognized research institutions, with a research project approved by an ethics committee for the protection of human subjects, will have access to the following data: the study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code. They can request access by emailing the principal investigator with all necessary information. After review, a data table will be sent.

REFERENCES:
- [Background] Gunning E, Uszynski MK. Effectiveness of the Proprioceptive Neuromuscular Facilitation Method on Gait Parameters in Patients With Stroke: A Systematic Review. Arch Phys Med Rehabil. 2019 May;100(5):980-986. doi: 10.1016/j.apmr.2018.11.020. Epub 2018 Dec 22. PMID 30582917
- [Background] Alexandre de Assis IS, Luvizutto GJ, Bruno ACM, Sande de Souza LAP. The Proprioceptive Neuromuscular Facilitation Concept in Parkinson Disease: A Systematic Review and Meta-Analysis. J Chiropr Med. 2020 Sep;19(3):181-187. doi: 10.1016/j.jcm.2020.07.003. Epub 2020 Dec 15. PMID 33362441
- [Background] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448